CLINICAL TRIAL: NCT05340218
Title: "Análisis Longitudinal Del Habla y Seguimiento a Corto Plazo de Las Facultades Cognitivas de Personas Mediante Una Serie de Pruebas: Lista de Palabras CERAD, Repite Los dígitos en Orden Inverso, TMTA-B, Prueba Del Reloj, Fluidez fonémica, comprensión Verbal Relaciones semánticas, y semánticas Alternas".
Brief Title: Short-term Automated Longitudinal Analysis of Speech and Language in Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Accexible (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18/475-E
Record Dates: First submitted 2022-03-29; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Speech analysis — Speech analysis to detect and monitor mild cognitive impairment

SUMMARY:
Validate speech analysis AI models:

* To contrast the accuracy of acceXible's platform as a screening tool in the detection of people with cognitive impairment and mild dementia.
* To evaluate the correlation between automatically analyzed linguistic variables and a combination of standard measures of cognition.
* To assess short-term variability in language ability among older adults, and to assess which aspects of language vary during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 55+ years of age with suspected MCI or diagnosis of dementia and obtains a score greater than 20 on the MMSE.
* Patients must have agreed to participate in the study and have voluntarily signed the informed consent.
* (Healthy) Participants without a diagnosis neurological, or psychiatric disorders. Or taking medication that can affect cognitive abilities.

Exclusion Criteria

* To have received a diagnosis of a significant psychiatric disorder or other cognitive impairment not due to neurodegeneration.
* To have significant vision problems that would affect the ability to perceive visual stimuli.
* To have significant hearing problems that would affect the ability to understand verbal cues.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-post variability of normal, MCI and dementia at both points of the study. | Change from the baseline cognitive function at 9 months.
  Through standard deviation of normal subjects, MCI and dementia, variations in language are measured by considering MMSE scores and the most significant variables of accexible's tests (image description test, phonetic verbal fluency test and semantic verbal fluency test).

SECONDARY OUTCOMES:
Correlation between cognitive tests and language variables obtained by the platform. | Every 6 to 9 months
  Correlation between: Standard measures of cognition (e.g., MMSE score) + behavioral and psychiatric symptoms of mild cognitive impairment and language.

OTHER OUTCOMES:
Accexible's model performance. | Every 6 to 9 months
  Percentage of patients classified correctly compared to the total number of sick patients, visualized at the ROC curve that allows to see the accuracy against the recall of the classifier. To contrast the accuracy of AcceXible's platform as a screening tool in the detection of people with cognitive impairment and mild dementia, a detection model has been developed from the analysis of the participants, acoustic, linguistic and semantic variables have been considered as well as audio characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Prevención de Deterioro Cognitivo, Madrid, Spain